CLINICAL TRIAL: NCT03389685
Title: Can Platelet Rich Plasma Reduce the Level of Pro-Inflammatory Synovial Fluid Biomarkers Following an Anterior Cruciate Ligament Tear
Brief Title: Can PRP Reduce Pro-Inflammatory Biomarkers Following ACL Injury
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID-19, Lack of Funding
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-02038
Record Dates: First submitted 2017-12-26; First posted 2018-01-03 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: ACL - Anterior Cruciate Ligament Rupture; ACL Injury
Keywords: Platelet Rich Plasma
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelet Rich Plasma (Experimental): Platelet Rich Plasma will be prepared using Genesis CS EmCyte PurePRP II system.
  Interventions: Biological: Platelet Rich Plasma
- Saline Placebo (Placebo Comparator): Unmarked syringe with 5 ml of saline
  Interventions: Other: Saline Placebo

INTERVENTIONS:
Biological: Platelet Rich Plasma — Pure PRPII®, leukocyte-poor, platelet rich plasma
  Arms: Platelet Rich Plasma
Other: Saline Placebo — saline solution
  Arms: Saline Placebo

SUMMARY:
The purpose of this single-center, double-blinded randomized control trial with prospective data collection is to assess the ability of platelet rich plasma (PRP) treatment to reduce the level of pro-inflammatory synovial fluid biomarkers following an acute anterior cruciate ligament (ACL) tear. The study will collect and analyze synovial fluid of patients presenting with an acute anterior cruciate ligament (ACL) tear with a second synovial fluid sampling at the time of surgery. It will compare synovial fluid biomarker levels between those receiving an intra-articular Platelet Rich Plasma (PRP) injection versus an intra-articular saline injection serving as a control. Post-operative clinical outcomes will also be assessed, including post-operative pain levels, incidence of post-operative knee stiffness and patient reported outcome scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients have suffered an acute ACL tear (initial presentation within 7 days of injury) with or without an associated meniscus injury
* Patient must undergo ACL reconstruction surgery

Exclusion Criteria:

* Mentally impaired (e.g, Alzheimer's subjects, dementia, etc.)
* Younger than 18 years of age
* Patients who have a multiligamentous injury
* Patients with underlying inflammatory arthropathies
* Previous ACL injury and/or reconstruction

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-09 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
synovial fluid biomarker levels | 2 Days
  The synovial fluid samples obtained at the two time points will be analyzed for the presence of 20 biomarkers using a multiplex bead assay (Milliplex®, Millipore, Billerica MA)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Strauss, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States